CLINICAL TRIAL: NCT05122273
Title: Assessment of the Effectiveness of Muscle Activating Training With the Use of EMG Biofeedback in Patients With Neuromuscular Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: EGZOTech (Industry)
Responsible Party: Sponsor
Other Study IDs: Orthos Trial
Record Dates: First submitted 2021-09-01; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Neuromuscular Diseases
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adults with confirmed neuromuscular disease: Children and adults with confirmed genetic Duchenne muscular dystrophy (DMD) or Becker muscular dystrophy (BMD), limb-girdle dystrophy, spinal muscular atrophy (SMA), myopathy or neuropathy.
  Interventions: Device: Stella BIO

INTERVENTIONS:
Device: Stella BIO — Individually planned therapeutic procedures, using, among others, the concept of EMG biofeedback

SUMMARY:
The aim of this study is to assess the impact of individually planned therapeutic procedures, using, among others, the concept of EMG biofeedback, to improve the general functional state, selected motor activities, stimulation and strength of specific muscle syndromes as well as postural parameters in children, adolescents and adults with neuromuscular diseases.

ELIGIBILITY:
Inclusion Criteria:

* confirmed genetic Duchenne muscular dystrophy (DMD) or Becker muscular dystrophy (BMD), limb-girdle dystrophy, spinal muscular atrophy (SMA), myopathy or neuropathy
* continued/uninterrupted rehabilitation process for 3 months
* patient's condition allowing full understanding of commands

Exclusion Criteria:

* patients using a respirator
* painful complaints
* after injuries and fractures in the last 6 months
* significant weakening of muscle strength, preventing movements and activation of selected muscle groups, visible in the EMG examination
* cognitive impairment-lack of or poor cooperation between the patient and the therapist,

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with confirmed genetic Duchenne muscular dystrophy (DMD) or Becker muscular dystrophy (BMD), limb-girdle dystrophy, spinal muscular atrophy (SMA), myopathy or neuropathy
Sampling Method: Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2021-11-20 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in functional assessment | baseline, after 12 weeks
  Motor Function Measure Scale Each MFM32 item is scored on a 4-point Likert scale from 0 (cannot initiate the task) to 3 (performs the task fully). Item scores are summed, and the raw score is transformed to an overall total score ranging from 0 (severe functional impairment) to 100 (no functional impairment).
Change in postural assessment by plurimeter (Rippstein) | baseline, after 12 weeks
  Spine curvature assessment in sagittal plane
Change in range of motion in upper and lower limb by goniometer | baseline, after 12 weeks
  Assessment of the changes in the range of motion in joints in the upper and lower limb measured by goniometer
Change in strength assessment | baseline, after 12 weeks
  Assessment of muscle strength using electrical dynamometer MicroFET2
Change in EMG assessment | baseline, after 12 weeks
  EMG assessment using Stella BIO device
Hammersmith Functional Motor Scale Expanded | baseline, after 12 weeks
  It contains 33 items which are scored on a scale of 0, 1, 2 with a total achievable score of 66.
  Score 2 = performs without modification/adaptation/compensation Score 1 = performs with modification/adaptation/compensation Score 0 = unable to perform A total score can be achieved by summing the scores for all the individual items. The total score can range from 0, if all the activities are failed, to 66, if all the activities are achieved.
North Star Ambulatory Assessment | baseline, after 12 weeks
  17-item rating scale that is used to measure functional motor abilities in ambulant children with Duchenne Muscular Dystrophy.
  The activities are graded as follows:
  2 - "Normal" - no obvious modification of activity
  1 - Modified method but achieves goal independent of physical assistance from another 0 - Unable to achieve independently This scale is ordinal with 34 as the maximum score indicating fully-independent function.
Change in postural assessment by scoliometer | baseline, after 12 weeks
  Assessment of the angle of the torso rotation in a sitting or standing position;
  Referral for scoliosis when rib slopeAngle of trunk rotation [ATR]is :
  8 degrees for underweight patients, 7 degrees for normal-weight patients, 6 degrees for overweight patients, and 5 degrees for obese patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Orthos, Warsaw, Poland